CLINICAL TRIAL: NCT06056050
Title: A Randomized, Blinded, Controlled Phase I Clinical Trial for Preliminary Evaluation of the Safety and Immunogenicity of Adsorbed Cell-free DPT Vaccine (for People Aged 6 Years and Above)
Brief Title: A Clinical Trial of Adsorbed Cell-free DPT Vaccine (5-component) (for People Aged 6 Years and Above)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: CanSino Biologics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CTP-Tdcp-001
Record Dates: First submitted 2023-09-19; First posted 2023-09-28 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2024-12

CONDITIONS: Diphtheria; Tetanus; Pertussis
Keywords: Vaccine; Five Components; Immunogenicity; Safety; ≥6 years; Acellular
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough | interventions — Tetanus Toxoid; Vaccines, Combined; Aging

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Experimental vaccine group 1A,≥18 years old (Experimental): 1 dose of Tdcp vaccine
  Interventions: Biological: Tetanus, Reduced Diphtheria and Acellular Pertussis (Five Components) Combined Vaccine, Adsorbed (Aged 6 Years and Older) (Tdcp)
- Control vaccine group 1B,≥18 years old (Active Comparator): 1 dose of PPV23 vaccine
  Interventions: Biological: 23-Valent Pneumococcal Polysaccharide Vaccine（PPV23）
- Experimental vaccine group 2A,12~17 years old (Experimental): 1 dose of Tdcp vaccine
  Interventions: Biological: Tetanus, Reduced Diphtheria and Acellular Pertussis (Five Components) Combined Vaccine, Adsorbed (Aged 6 Years and Older) (Tdcp)
- Control vaccine group 2B,12~17 years old (Active Comparator): 1 dose of PPV23 vaccine
  Interventions: Biological: 23-Valent Pneumococcal Polysaccharide Vaccine（PPV23）
- Experimental vaccine group 3A,6~11 years old (Experimental): 1 dose of Tdcp vaccine
  Interventions: Biological: Tetanus, Reduced Diphtheria and Acellular Pertussis (Five Components) Combined Vaccine, Adsorbed (Aged 6 Years and Older) (Tdcp)
- Control vaccine group 3B,6~11 years old (Active Comparator): 1 dose of DT vaccine
  Interventions: Biological: Diphtheria and Tetanus Combined Vaccine, Adsorbed (DT)

INTERVENTIONS:
Biological: Tetanus, Reduced Diphtheria and Acellular Pertussis (Five Components) Combined Vaccine, Adsorbed (Aged 6 Years and Older) (Tdcp) — 1 dose of Tdcp vaccine (0.5ml) on Day 0
  Arms: Experimental vaccine group 1A,≥18 years old; Experimental vaccine group 2A,12~17 years old; Experimental vaccine group 3A,6~11 years old
Biological: 23-Valent Pneumococcal Polysaccharide Vaccine（PPV23） — 1 dose of PPV23 vaccine (0.5ml) on Day 0
  Arms: Control vaccine group 1B,≥18 years old; Control vaccine group 2B,12~17 years old
Biological: Diphtheria and Tetanus Combined Vaccine, Adsorbed (DT) — 1 dose of DT vaccine (0.5ml) on Day 0
  Arms: Control vaccine group 3B,6~11 years old

SUMMARY:
Pertussis is an acute respiratory infectious disease caused by Bordetella pertussis, diphtheria is an acute upper respiratory infectious disease caused by Gram-positive Corynebacterium diphtheriae, and tetanus is a highly fatal disease caused by Clostridium tetani infection. Currently, there is no clinical trial registration of Diphtheria, tetanus, and pertussis (DPT) vaccine applicable to ≥6 years of age in China, therefore, the five-component acellular DPT combination vaccine developed by our research has a promising future.

DETAILED DESCRIPTION:
The vaccines used in China's immunization program for the prevention of pertussis, tetanus and diphtheria include the adsorbed cell-free diphtheria-tetanus-acellular pertussis vaccine (DTaP) and the diphtheria-tetanus-acellular tetanus vaccine (DT) and tetanus vaccine. Among them, DTaP vaccination is for children from 3 months of age to 6 years of age, with one dose each at 3, 4, 5, and 18 months of age; DT vaccination is for children under 12 years of age, with one dose at 6 weeks of age after completing four doses of DTaP vaccination. However, infant and young child vaccination is no longer sufficient to prevent the threat of this disease, mainly due to the rapid decay of immune protection in adolescents and adults, and infections in this population, which are the main source of infection leading to infection in infants and young children, have been a number of new preventive strategies are being evaluated.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 6 years of age.
* Willingness to provide proof of identity.
* The informed consent of the volunteer and/or the guardian and/or the delegate must be obtained and the informed consent form must be signed.
* Volunteers are able and willing to comply with the requirements of the clinical trial protocol and are able to complete the full study follow up.
* Volunteers aged 6-11 years who have completed 4 doses of DPT-containing vaccine, but have not received the 5th dose, and have ≥3 years between the 4th dose.
* Volunteers aged ≥12 years must not have received any of the components of the DPT-containing vaccine within 5 years.

Exclusion Criteria:

* Persons with fever prior to vaccination, with axillary temperature > 37.0°C.
* A female with a positive urine pregnancy test or a breastfeeding volunteer, where the volunteer or her partner has a plan to become pregnant within 180 days.
* Adults with severe cardiovascular disease, hypertension (systolic blood pressure ≥160mmHg, diastolic blood pressure ≥100mmHg) that cannot be controlled by medication, or other severe chronic diseases.
* Abnormal and clinically significant results of preimmunization blood tests, blood biochemistry and urine tests.
* Persons who have suffered from one of the diseases of diphtheria or tetanus, or who have suffered from whooping cough in the last three years.
* Volunteers ≥12 years of age who have received pneumococcal polysaccharide/conjugate-containing vaccine within 4 years.
* Individuals who have had household contact with individuals diagnosed with pertussis, diphtheria, tetanus in the past 30 days.
* Individuals who are allergic to the components of the study vaccine or who have developed an allergy during previous administration of the same vaccine; individuals with a previous history of severe allergies, such as urticaria, anaphylaxis, respiratory distress, angioneurotic edema, or asthma.
* History of convulsions, epilepsy, encephalopathy and serious neurological disorders (e.g., transverse myelitis, Guillain-Barre syndrome, demyelinating diseases, etc.), etc.
* Individuals with primary and secondary immune impairment (history of thyroid, pancreas, liver, spleen, kidney disease or removal, or need for treatment due to thyroid disease within the past 12 months), who have received immunosuppressive therapy within 3 months.
* Physician-diagnosed coagulation abnormalities (e.g., coagulation factor deficiencies, coagulopathies, platelet abnormalities) or significant bruising or coagulation disorders.
* Persons with acute febrile illnesses and current patients with infectious diseases who have had a history of moderately high fever (axillary temperature ≥38.0°C) or cardiopulmonary disease (frequent asthma attacks) within the past 3 days.
* Has received another investigational drug or vaccine within 1 month prior to receiving the experimental drug, or is planning to participate or is participating in a clinical study of any other drug.
* Received live attenuated vaccine within 14 days prior to receiving the test drug and subunit vaccine or inactivated vaccine within 7 days prior to receiving the test drug.
* Any other factors that, in the judgment of the investigator, make the volunteer unsuitable for participation in a clinical trial.

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-12-06 (Actual); Primary Completion 2024-04-13 (Actual); Study Completion 2025-09-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse reactions 0-30 days after vaccination | 0-30 days after vaccination

SECONDARY OUTCOMES:
Incidence of adverse reactions within 30 minutes of vaccination | Within 30 minutes of vaccination
Incidence of adverse reactions/adverse events 0-7 days after vaccination | 0-7 days after vaccination
Incidence of adverse events 0-30 days after vaccination | 0-30 days after vaccination
Incidence of severe adverse events (SAE) 360 days after vaccination in the 6-11 years old group | 360 days after vaccination
Incidence of SAE 180 days after vaccination in the 12-17 year old group and the ≥18 years old group | 180 days after vaccination
Hemoglobin content (HGB) on day 4 after vaccination | Day 4 after vaccination
White blood cell count on day 4 after vaccination | Day 4 after vaccination
Alanine aminotransferase (ALT) in blood on day 4 after vaccination | Day 4 after vaccination
Aspartate aminotransferase (AST) in blood on day 4 after vaccination | Day 4 after vaccination
Total bilirubin (TBIL) in blood on day 4 after vaccination | Day 4 after vaccination
Protein in urine on day 4 after vaccination | Day 4 after vaccination
Erythrocytes in urine on day 4 after vaccination | Day 4 after vaccination
Antibody Positive Turnover of Serum Anti-Diphtheria Toxoid(DT), Tetanus Toxoid(TT), Pertussis Toxoid(PT), Filamentous hemagglutmin(FHA), Pertactin(PRN), FIM bridal agglutinogens(FIM) 2&3 at 30 days after vaccination | 30 days after vaccination
Antibody Positivity of Serum Anti-DT, TT, PT, FHA, PRN, FIM 2&3 at 30 days after vaccination | 30 days after vaccination
Geometric Mean Concentration (GMC) of Serum Anti-DT, TT, PT, FHA, PRN, FIM 2&3 at 30 days after vaccination | 30 days after vaccination
Proportion of serum anti-PRN, FIM 2&3 antibodies ≥5, 10, 20 IU/ml 30 days after vaccination | 30 days after vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Shaanxi Center for Disease Control and Prevention, Xi'an, Shaanxi, China

REFERENCES:
- [Derived] Liu X, Wei C, Huang H, Wan J, Li Y, Wang F, Li S, Wang Y, Wang X, Wang X, Sui X, Gou J, Zhu T, Ma X, Hu W. Preliminarily evaluation the safety and immunogenicity of tetanus, reduced diphtheria and acellular pertussis (five components) combined vaccine, adsorbed (Tdcp) in participants aged 6 years and above: a blinded and randomised, and controlled phase I clinical trial. Front Immunol. 2025 Sep 5;16:1616574. doi: 10.3389/fimmu.2025.1616574. eCollection 2025. PMID 40977696